CLINICAL TRIAL: NCT00991614
Title: Treatment of Duodenal or Gastric Outlet Obstruction and Duodenal Strictures Caused by Malignant Neoplasms With the EVOLUTION® Duodenal Stent
Brief Title: EVOLUTION® Duodenal Stent for Duodenal or Gastric Outlet Obstruction Caused by Malignant Neoplasms
Status: Completed | Type: Observational
Sponsor: Cook Group Incorporated (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-005
Record Dates: First submitted 2009-08-13; First posted 2009-10-08 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Duodenal Obstruction; Gastric Outlet Obstruction
MeSH Terms: conditions — Duodenal Obstruction; Gastric Outlet Obstruction

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- EVOLUTION® Duodenal Stent
  Interventions: Device: EVOLUTION® Duodenal Stent

INTERVENTIONS:
Device: EVOLUTION® Duodenal Stent — EVOLUTION® Duodenal Stent
  Other Names: TC325

SUMMARY:
The objective of this investigation is to compile clinical experience on the use of the Evolution® Duodenal Stent (Cook Ireland), a CE marked device intended for the palliative treatment of duodenal or gastric outlet obstruction and duodenal strictures caused by malignant neoplasms. It is not the goal to change the usual treatment practice of the investigator or the center, nor to collect information on uses outside the product's indications. Patients will be treated as per usual medical practices.

ELIGIBILITY:
Inclusion Criteria:

* Patients for whom this device would be chosen in standard practice

Exclusion Criteria:

* Patients for whom this device would not normally be chosen in standard practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are referred into regional specialty centers for treatment of GI malignancy.
Sampling Method: Non-Probability Sample
Enrollment: 110 (Actual)
Dates: Start 2009-12; Primary Completion 2011-06 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Patency of the stent | 14 days

SECONDARY OUTCOMES:
Procedural success, implant duration, symptom resolution | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Professor Guido Costamagna, MD, Principal Investigator — U.O. Endoscopia Digestiva Chirurgica
Locations (6):
- Westmead Hospital, Sydney, Australia
- Hopital Saint-Luc / CHUM, Montreal, Quebec, Canada
- Institution for Clinical and Experimental Medicine, Prague, Czechia
- Italy (2):
  - IRCCS Instituto Clinico Humanitas, Milan
  - U.O. Endoscopia Digestiva Chirurgica, Rome
- Erasmus MC University Medical Center, Rotterdam, Netherlands

REFERENCES:
- [Derived] Tringali A, Didden P, Repici A, Spaander M, Bourke MJ, Williams SJ, Spicak J, Drastich P, Mutignani M, Perri V, Roy A, Johnston K, Costamagna G. Endoscopic treatment of malignant gastric and duodenal strictures: a prospective, multicenter study. Gastrointest Endosc. 2014 Jan;79(1):66-75. doi: 10.1016/j.gie.2013.06.032. Epub 2013 Aug 6. PMID 23932009